CLINICAL TRIAL: NCT02233803
Title: A Randomised, Multi-centre, Open Label, Cross-over Non-inferiority Study to Evaluate Efficacy, Safety and Tolerability of Neumoterol 400 and Symbicort Forte in Adults With Asthma
Brief Title: A Non-inferiority Study to Evaluate Efficacy, Safety and Tolerability of NEUMOTEROL® 400 and SYMBICORT® Forte in Adults With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201435
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: tolerability; NEUMOTEROL; efficacy; budesonide/formoterol fumarate 400/12 mcg; safety; Asthma; pharmacodynamics
MeSH Terms: conditions — Asthma | interventions — Single Person; Nebulizers and Vaporizers; Budesonide; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1: BFF 400/12mcg to BFF 320/9mcg (Experimental): Subjects will receive Regimen A in Treatment Period 1 followed by Regimen B in Treatment Period 2. The treatment periods will be separated by a wash out period of 4 weeks. Regimen A: Subjects will be instructed to take each morning and evening, 1 inhalation from a single capsule containing BFF (400/12 mcg) by single capsule inhaler. Regimen B: Subjects will be instructed to take each morning and evening,1 inhalation from BFF (320/9 mcg) TURBUHALER inhaler.
  Interventions: Drug: NEUMOTEROL 400 (BFF 400/12 mcg) single capsule inhaler; Drug: SYMBICORT forte (BFF 320/9mcg) TURBUHALER inhaler; Drug: NEUMOTEX 400 (Budesonide 400 mcg); Drug: Salbutamol 100 mcg pMDI
- Sequence 2: BFF 320/9mcg to BFF 400/12mcg (Experimental): Subjects will receive Regimen B in Treatment Period 1 followed by Regimen A in Treatment Period 2. The treatment periods will be separated by a wash out period of 4 weeks. Regimen A: Subjects will be instructed to take each morning and evening, 1 inhalation from a single capsule containing BFF (400/12 mcg) by single capsule inhaler. Regimen B: Subjects will be instructed to take each morning and evening,1 inhalation from BFF (320/9 mcg) TURBUHALER inhaler.
  Interventions: Drug: NEUMOTEROL 400 (BFF 400/12 mcg) single capsule inhaler; Drug: SYMBICORT forte (BFF 320/9mcg) TURBUHALER inhaler; Drug: NEUMOTEX 400 (Budesonide 400 mcg); Drug: Salbutamol 100 mcg pMDI

INTERVENTIONS:
Drug: NEUMOTEROL 400 (BFF 400/12 mcg) single capsule inhaler — Micronized 400 mcg budesonide+ 12 mcg formoterol fumarate along with micronized and crystalline lactose monohydrate (excipient), per capsule dispensed by single capsule inhaler, twice daily (administered once in the morning and once in the evening approximately 12 hours later).
Drug: SYMBICORT forte (BFF 320/9mcg) TURBUHALER inhaler — Unit dose containing 320 mcg budesonide and 9 mcg formoterol fumarate (as dihidrate) along with lactose monohydrate as excipient. Administered as inhalation by TURBUHALER inhaler, twice daily (once in the morning and once in the evening approximately 12 hours later)
Drug: NEUMOTEX 400 (Budesonide 400 mcg) — Budesonide 400mcg will be administered to all the subjects twice daily, during the Run-in and Washout Periods
Drug: Salbutamol 100 mcg pMDI — Salbutamol 100mcg will be administered as pMDI on demand, as rescue medication, throughout the entire study period until Visit 5

SUMMARY:
This Phase IV study is an a multi-centre, randomised open label, two way cross-over design to evaluate the efficacy, safety, and tolerability of NEUMOTEROL 400 in subjects with asthma. The study will be used to demonstrate the non-inferiority of Budesonide/Formoterol Fumarate combination (BFF) 400/12 micrograms (mcg) single capsule inhaler (NEUMOTEROL 400) compared with BFF 320/9 mcg SYMBICORT Forte TURBUHALER® inhaler.

The population for this study will be adult subjects (>=18 and <=80 years) with a diagnosis of asthma who have a pre-bronchodilator forced expiratory volume in one second (FEV1) of 40% to 85% of the predicted normal value, and are receiving a stable dose of inhaled corticosteroid inhaled corticosteroid (ICS) with or without long-acting beta-adrenergic agonist (LABA) prior to screening.

The study will consist of six phases: Prescreening, Screening/Run-in (4 weeks), Treatment Period 1 (4 weeks), Washout (minimum 4 weeks), Treatment Period 2 (4 weeks) and Follow-up (1 week). The total duration of the study for each subject will be at least 17 weeks. There will be up to 6 study visits and a follow-up telephone call.

Pre-screening Visit will allow subjects who had recent asthma medication changes to be stabilized prior to Screening. During the run-in and wash-out periods, all the subjects will receive budesonide dry powder inhaler (DPI) 400 mcg twice daily (BID) (NEUMOTEX™ 400) and salbutamol 100mcg pressurized metered dose inhaler (pMDI) on demand, as rescue medication. The dose of NEUMOTEROL 400 (400/12 mcg) and SYMBICORT Forte (320/9 mcg) will be one inhalation BID, and each treatment will be given to all subjects for 4 weeks (with a 4-week Washout Period between treatments).

The study will include 300 subjects for screening so that at least 210 will be randomised and a minimum of 168 subjects complete the study/are evaluable. Half the subjects will be on Regimen A in Treatment Period 1and will then be crossed over to Regimen B in Treatment Period 2, and vice versa. Regimen A: BFF (400/12 mcg) by single capsule inhaler. Regimen B: BFF (320/9 mcg) TURBUHALER inhaler. The treatment periods will be separated by a washout Period of 4 weeks.

NEUMOTEROL and NEUMOTEX are trademarks of the GSK group of companies SYMBICORT and TURBUHALER are trademarks of AstraZeneca

ELIGIBILITY:
Inclusion Criteria:

* Male or female >=18 and <=80 years of age with a diagnosis of asthma at the time of signing the informed consent
* A female subject is eligible to participate if she is of: Non-child bearing potential defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone >40 milli-international unit/milliliter (mIU/mL) and oestradiol <40 picogram/millilitre (pg/mL) [<147 picomol/litre] is confirmatory) ; Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study from Screening to follow-up contact) if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrolment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. After confirmation of their postmenopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential and is abstinent or agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) before the start of dosing to sufficiently minimise the risk of pregnancy at that point. Female subjects must agree to use contraception until at least 2 days post the last dose of study treatment ; Abstinence from penile-vaginal intercourse must be consistent with the preferred and usual lifestyle of the subject
* Severity of disease: A best pre-bronchodilator FEV1 of >=40% to <=85% of the predicted normal value at Visit 1 (Screening and Run-in Visit). . Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations.
* Reversibility of disease: Demonstrated >=12% and >=200 mL reversibility of FEV1 within 10 to 40 minutes after 2 to 4 inhalations of salbutamol inhalation aerosol (or equivalent nebulised treatment with salbutamol solution) at Visit 1 (Screening and Run-in Visit)
* Current anti-asthma therapy: All subjects must be using an ICS with or without LABA for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). Two populations are eligible for enrolment: Subjects maintained on ICS monotherapy (Budesonide 400 mcg to 800 mcg BID or equivalent) for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit) or Subjects maintained on an ICS/LABA combination product (e.g., NEUMOTEROL 200/6 BID or 400/12 mcg BID or equivalent by other combination products or by separate inhalers) for at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). Subjects taking budesonide/formoterol as needed must switch to maintenance dosing (excluding the highest dose) with use of a SABA for symptom relief at least 8 weeks and a stable dose for at least 4 weeks before Visit 1 (Screening and Run-in Visit). NOTE: Subjects on low dose ICS monotherapy should only be enrolled, if, in the opinion of the investigator, after review of their medical history and clinical examination, they will be able to benefit from both an increase in ICS dose and the addition of LABA therapy arising from and ICS/LABA combination
* Ability to withhold LABA therapy : Other than what is provided during the study, LABA therapy is not permitted on the day of Visit 1(Screening and Run-in Visit) and throughout the entire study. The last dose of pre-study LABA and LABA/ICS combinations are to be taken on the day before Visit 1. According to investigators judgement, patients should be able to withhold LABA therapy during the run-in and wash-out period.
* SABA: All subjects must be able to replace their current SABA treatment with rescue salbutamol at Visit 1 (Screening and Run-in Visit) for use as needed for the duration of the study. Subjects must be able to withhold salbutamol for at least 6 hours before each study visit
* Liver safety criteria: Alanine aminotransferase (ALT) <=2×the upper limit of normal (ULN), Alkaline phosphatase and bilirubin <=1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%) at Visit 1 (Screening and Run-in Visit)
* Electrocardiography (ECG) safety criteria : The subject must have no ECG abnormalities that would, in the opinion of investigator, compromise subject safety, or significantly affect subject's ability to complete the trial. As such, the investigator will determine the clinical significance of any ECG abnormality and determine if a subject is precluded from entering the study. At Visit 1 (Screening and Run-in Visit), ECG safety criteria must be: QT interval corrected for heart rate (QTc) <450 microseconds (msec) or QTc <480 msec for patients with bundle branch block. The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. The QTc should be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period. Investigators will be responsible for ensuring appropriate clinical interpretation of ECGs.
* The subject and/or the subject's legal guardian (if applicable) must be capable of giving informed consent/assent, which includes compliance with the study requirements and restrictions listed in the consent/assent form

Exclusion Criteria:

* History of life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 10 years
* Respiratory infection: Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Visit 1 (Screening and Run-in Visit) and led to a change in asthma management, or in the opinion of the investigator, is expected to affect the subject's asthma status or ability to participate in the study
* Asthma exacerbation: Any asthma exacerbation requiring oral corticosteroids within 12 weeks of Visit 1 (Screening and Run-in Visit)or that resulted in overnight hospitalisation requiring additional treatment for asthma within 6 months before Visit 1 (Screening and Run-in Visit)
* Asthma severely uncontrolled: ACT bellow 15 at Visit 1
* Concurrent respiratory disease: A subject must not have current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease (COPD), or other respiratory abnormalities other than asthma
* Other concurrent diseases/abnormalities: A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study. Additional excluded conditions/diseases may include (but not limited to): congestive heart failure, known aortic aneurysm, clinically significant coronary heart disease, clinically significant cardiac arrhythmia, stroke within 3 months of Visit 1 (Screening and Run-in Visit), uncontrolled hypertension (two or more measurements with systolic blood pressure [BP] >160 millimeter mercury [mmHg], or diastolic BP >100 mmHg), Recent or poorly controlled peptic ulcer, Haematologic, hepatic, or renal disease, Immunologic compromise, Current malignancy(History of malignancy is acceptable only if subject has been in remission for one year before Visit 1 (Screening and Run-in Visit) (remission = no current evidence of malignancy and no treatment for the malignancy in the 12 months before Visit 1 [Screening and Run-in Visit]), Tuberculosis (current or untreated) (subjects with a history of tuberculosis infection who have completed an appropriate course of anti-tuberculous treatment may be suitable for study entry provided that there is no clinical suspicion of active or recurrent disease), Cushing's disease, Addison's disease, uncontrolled diabetes mellitus, uncontrolled thyroid disorder and recent history of drug or alcohol abuse.
* Evidence of a severe exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalisation or emergency department visit due to asthma that required systemic corticosteroids between Visit 1 (Screening and Run-in Visit) and Visit 2 (randomization and Treatment Period 1 Baseline Visit)
* Oropharyngeal examination: A subject will not be eligible for the Run-in if he/she has clinical visual evidence of candidiasis at Visit 1(Screening and Run-in Visit)
* Investigational medications: A subject must not have administered any investigational drug within 30 days before Visit 1(Screening and Run-in Visit) or within five half-lives of the prior investigational drug (whichever is the longer of the two). The prior investigational drug half-life may be confirmed with the prior investigational study sponsor or by consulting relevant study documentation
* Allergies: Drug allergy: Any adverse reaction including immediate or delayed hypersensitivity to any beta2 agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the BFF TURBUHALER inhaler and capsules (i.e., lactose) ; Milk protein allergy: history of severe milk protein allergy
* Concomitant medications: Administration of prescription or over the counter medication that would significantly affect the course of asthma, or interact with study treatment, such as: anticonvulsants (barbiturates, hydantoins, carbamazepine); polycyclic antidepressants; beta-adrenergic blocking agents; phenothiazines; and monoamine oxidase (MAO) inhibitors; Immunosuppressive medications: A subject must not be using or require use of immunosuppressive medications during the study; cytochrome P450 3A4 (CYP3A4) inhibitors: Subjects who have received a potent CYP3A4 inhibitor within 4 weeks of Visit 1(Screening and Run-in Visit) (e.g., ritonavir, ketoconazole, itraconazole) ; Unable to refrain from the use of prescription or nonprescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) before the first dose of study treatment, unless in the opinion of the investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety; Any subjects that have previously received or are currently receiving omalizumab .
* Medications prior to Screening : Use of the following medications within the defined times prior to Visit 1 (Screening and Run-in Visit): Corticosteroids (Systemic, oral, or depot corticosteroids) (12 Weeks); inhaled corticosteroids(Monotherapy or in combination with a LABA for a minimum of 8 weeks and maintained on a stable dose for 4 weeks prior to Visit 1); SABA(6 hours prior to all spirometry assessments) (Study supplied SABA is permitted); LABA (Oral LABAs, inhaled LABAs or combination products containing inhaled LABAs) (1 day); Theophylline, ketotifen, sodium cromoglycate, nedocromil sodium (1 day); Short-acting anti-muscarinics (12 hours), Long-acting anti-muscarinics (7 days), Potent cytochrome P450 3A4 inhibitors (4 weeks), Leukotriene modifiers (48 hours), Immunosuppressive medication (6 months), Anti- immunoglobulin E (12 weeks); Prescription or over the counter medication that would significantly affect the course of asthma, or interact with sympathomimetic amines such as: anticonvulsants (1 day); Herbal medicines (Prescription or nonprescription drugs, including vitamins, herbal and dietary supplements [including St John's worth] unless in the opinion of the investigator and medical monitor the medication will not interfere with the study procedures or compromise subject safety) (7 days [or 14 days if the drug is a potential enzyme inducer] or five half-lives [whichever is longer]); Chinese traditional medicines (1 day) ; Any other investigational drug (30 days or within five half-lives, whichever is longer).
* Compliance: A subject will not be eligible if he/she or his/her parent or legal guardian has any infirmity, disability, disease, or geographical location that seems likely (in the opinion of the investigator) to impair compliance with any aspect of this study protocol, including visit schedule and completion of the daily diaries
* Tobacco use: Current smoker or a smoking history of >=10 pack-years (e.g., 20 cigarettes/day for 10 years). A subject must not have used inhaled tobacco products within the past 3 months (e.g., cigarettes, cigars or pipe tobacco). One pack year is defined as 20 manufactured cigarettes (1 pack) smoked per day for 1 year.
* Pregnant females as determined by urine test at Visit 1 (Screening and Run-in Visit) or pre-dosing. A confirmatory serum pregnancy test is required if the urine test is questionable or positive
* Lactating females
* A positive hepatitis B surface antigen or positive hepatitis C test result
* Subject is mentally or legally incapacitated Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Argentina (10):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Vicente López, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Berazategui, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Monte Grande
  - GSK Investigational Site, Rosario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in adult asthma participants, at 11 centres in Argentina from 14 November 2014 to 11 December 2015.
Pre-assignment Details: Total 6 phases of study; pre-screening, screening/run-in, treatment period (TP) 1 washout, TP2, and follow-up. Out of total 239 enrolled participants, only 199 participants were randomized. 29 were screen failures and 10 were Run-in failures. One participant not randomized as the target number of participants for study was reached
Groups:
- NEUMOTEROL 400/ SYMBICORT FORTE: During TP1, participants received Regimen A where the eligible participants received, 1 inhalation of budesonide/formoterol fumarate (BFF), 400/12 microgram [mcg] (NEUMOTEROL 400) by single capsule inhaler each morning and evening for 4- weeks (Wks). This was followed by a wash out period of 4 Wks , during which all the participants received budesonide DPI 400 mcg (NEUMOTEX 400) twice daily. The wash-out period was followed by Regimen B during which the eligible participants took, 1 inhalation of BFF 320/9 mcg (SYMBICORT FORTE), by turbuhaler inhaler each morning and evening, for 4-Wks. Additionally all participants were allowed to take rescue medication (salbutamol 100 mcg) during the study.
- SYMBICORT FORTE/ NEUMOTEROL 400: During TP1, the participants received Regimen B where the eligible participants took, 1 inhalation of BFF 320/9 mcg (SYMBICORT FORTE), by turbuhaler inhaler each morning and evening for 4-Wks. This was followed by a wash out period of 4 Wks, during which all the participants received budesonide DPI 400 mcg (NEUMOTEX 400) twice daily. It was then followed by Regimen A during which eligible participants received, 1 inhalation of NEUMOTEROL 400 by single capsule inhaler each morning and evening, for 4-Wks. Additionally all participants were allowed to take rescue medication (salbutamol 100 mcg) during the study.
Period: Treatment Period 1 (4-Wks)
Arm/Group | NEUMOTEROL 400/ SYMBICORT FORTE | SYMBICORT FORTE/ NEUMOTEROL 400
Started | 100 | 99
Completed | 97 | 95
Not Completed | 3 | 4
Not completed — Protocol-defined stopping criteria reach | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period (4-Wks)
Arm/Group | NEUMOTEROL 400/ SYMBICORT FORTE | SYMBICORT FORTE/ NEUMOTEROL 400
Started | 97 | 95
Completed | 95 | 93
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Treatment Period 2 (4-Wks)
Arm/Group | NEUMOTEROL 400/ SYMBICORT FORTE | SYMBICORT FORTE/ NEUMOTEROL 400
Started | 95 | 93
Completed | 93 | 91
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: The eligible participants were randomised to receive either Regimen A in TP1 and Regimen B in TP2, or Regimen B in TP1 and Regimen A in TP2 according to the randomisation schedule. Both the TPs were separated by a wash out period of 4 weeks. Regimen A: 1 inhalation of budesonide/formoterol fumarate (BFF), 400/12 microgram [mcg] (NEUMOTEROL 400) by single capsule inhaler each morning and evening. Regimen B: 1 inhalation of BFF 320/9 mcg (SYMBICORT FORTE) by turbuhaler inhaler each morning and evening. Additionally all participants were allowed to take rescue medication (salbutamol 100 mcg) during the study.
Arm/Group | Total
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 57
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European Heritage | 199

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Morning Forced Expiratory Volume in One Second (FEV1) at Day (D)29
Description: FEV1 is maximal amount of air, forcefully exhaled in one second. Trough FEV1 is defined as morning prebronchodilator and predose: 12 hours (h) after last evening dose D28 at end of each TP. Measured by spirometer in morning, before using bronchodilator and pre-dosing at wk1 D1 and wk4 D29 of each TP and test was performed within 30 minutes prior to dosing. Change from BL was analysed using mixed effects ANCOVA model fitting terms for subject-level (SL) BL, Adjusted period-specific (PS) BL, treatment group and period, with participant as random effect. PS BL value is pre-dose assessment collected on D1 of each TP. SL BL is arithmetic mean of PS BL values of participant. If only one of PS BL value is missing for participant, SL BL took value of other BL. If both PS BL values were missing, SL BL was set to missing. Period level BL=PS BL - associated SL BL.
Time Frame: BL (D1) and D29 (each TP)
Population: The intent to treat (ITT) population comprised of all randomized participants who received at least one dose of study treatment. This population was based on the treatment to which the participant was randomized. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Groups:
- NEUMOTEROL 400: Eligible participants received NEUMOTEROL 400 during TP1 or TP2 as per their randomization. The TPs were separated by washout period of 4-wks during which participants received NEUMOTEX 400, twice daily. The participants were allowed to take salbutamol 100mcg pressurized metered dose inhaler (pMDI), as rescue medication.
- SYMBICORT FORTE: Eligible participants received Symbicort forte during TP1 or TP2 as per their randomization . The TPs were separated by washout period of 4-wks during which participants received NEUMOTEX 400, twice daily. The participants were allowed to take salbutamol 100mcg pMDI, as rescue medication.
Arm/Group | NEUMOTEROL 400 | SYMBICORT FORTE
Number analyzed (Participants) | 188 | 188
Litre (L) | 0.194 (0.0213) | 0.150 (0.0213)
Statistical Analysis 1: Comparison: NEUMOTEROL 400 vs SYMBICORT FORTE; Sample size calculations are based on the primary efficacy endpoint (change from baseline in trough FEV1 at day 29). Assuming a within-subject standard deviation of 210 mL, 168 completed subjects are required to demonstrate the non-inferiority of BFF 400/12 mcg SINGLE CAPSULE INHALER and BFF 320/9 mcg TURBUHALER BID, assuming a true difference of -50 mL with 90% power and a 2.5% one-sided significance level. The pre-specified NI margin is set at -1.25mL; Test type: Non-Inferiority or Equivalence — Non-inferiority (NI) is demonstrated as the lower limit of CI for the difference is greater than the pre-specified NI margin of -1.25ML. The lower limit of the 95% CI for the treatment difference (NEUMOTEROL 400 -Symbicort Forte) was greater than the pre-specified non-inferiority margin of -1.25 mL; Difference of LS means = 0.044, 95% CI 2-sided [-0.008 to 0.096]

2. Secondary Outcome: FEV1 Area Under the Curve (AUC) (0-10 h) at D1 of Each TP
Description: FEV1 is the maximal amount of air that can be forcefully exhaled in one second. FEV1 AUC (0 to 10h) was measured at beginning of each TP. AUC was derived using values observed at the following timepoints: 0 minute (pre-morning dosing), 5 minutes (m), 15m, 30m, 1, 2, 5, and 10h; post morning dosing FEV1 values on D1 of each TP. Pre-dose was taken as, 0h timepoint on the visit of interest, and all subsequent timepoints were calculated relative to that timepoint. FEV1 AUC was analysed using mixed effects ANCOVA model fitting terms for subject-level (SL) BL, Adjusted period-specific(PS) BL, treatment group and period, with participant as random effect.
Time Frame: (0-10 h) at D1 (each TP)
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L*hrs
Groups:
- NEUMOTEROL 400: Eligible participants received NEUMOTEROL 400 during TP1 or TP2 as per their randomization. The TPs were separated by washout period of 4-wks during which participants received NEUMOTEX 400, twice daily. The participants were allowed to take salbutamol 100mcg pMDI, as rescue medication.
- SYMBICORT FORTE: Eligible participants received Symbicort forte during TP1 or TP2 as per their randomization. The TPs were separated by washout period of 4-wks during which participants received NEUMOTEX 400, twice daily. The participants were allowed to take salbutamol 100mcg pMDI, as rescue medication.
Arm/Group | NEUMOTEROL 400 | SYMBICORT FORTE
Number analyzed (Participants) | 193 | 194
L*hrs | 24.573 (0.1840) | 23.593 (0.1836)
Statistical Analysis 1: Comparison: NEUMOTEROL 400 vs SYMBICORT FORTE; Test type: Superiority or Other; Difference of LS means = 0.980, 95% CI 2-sided [0.576 to 1.384]

3. Secondary Outcome: Change From BL in Asthma Control Test (ACT) at 4 Wks for Each TP
Description: ACT was basically a five item questionnaire, to measure participant's asthma control. It comprised of five possible answers to each question, associated with a score of 1 to 5 (1=poor control and 5=good control), wherein the scores from each question were summed to give an overall score (5=poor control and 25=complete control). ACT was recommended during each visit and was completed by the participant before any procedures were performed, avoiding any influence of the participants response. Change from BL was analysed using mixed effects ANCOVA model fitting terms for subject-level (SL) BL, Adjusted period-specific(PS) BL, treatment group and period, with participant as random effect. PS BL value, is pre-dose assessment collected on D1 of each TP. SL BL, is arithmetic mean of PS BL values of participant. Participants with an ACT below 15 were excluded from the study.
Time Frame: BL up to W4 (each TP)
Population: ITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | NEUMOTEROL 400 | SYMBICORT FORTE
Number analyzed (Participants) | 188 | 188
units on scale | 1.6 (0.20) | 1.0 (0.20)
Statistical Analysis 1: Comparison: NEUMOTEROL 400 vs SYMBICORT FORTE; Test type: Superiority or Other; Difference of LS means = 0.6, 95% CI 2-sided [0.1 to 1.1]

ADVERSE EVENTS:
Time Frame: Up to 14 wks
Description: Safety population comprised of all participants who received at least one dose of study treatment. This population was based on the treatment the participant actually received.
Arm/Group | NEUMOTEROL 400 | SYMBICORT FORTE
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/194
Serious Adverse Events (participants affected / at risk) | 1/193 | 1/194
Other Adverse Events (participants affected / at risk) | 10/193 | 11/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEUMOTEROL 400 (N=193) | SYMBICORT FORTE (N=194)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEUMOTEROL 400 (N=193) | SYMBICORT FORTE (N=194)
Headache (Nervous system disorders) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.